CLINICAL TRIAL: NCT02923648
Title: Lung Obstruction in Adulthood of Prematurely Born (LUNAPRE)
Acronym: LUNAPRE
Status: Active, not recruiting | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Swedish Heart Lung Foundation (Other); The Swedish Research Council (Other Government); Region Stockholm (Other Government); Stockholm South General Hospital (Other); University of California, San Francisco (Other); Kyoto University (Other); Göteborg University (Other); University of Oulu (Other)
Responsible Party: Principal Investigator, Asa Wheelock, Associate professor, Karolinska Institutet
Other Study IDs: 2012/1872-31/4
Record Dates: First submitted 2016-10-03; First posted 2016-10-04 (Estimated); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Premature Birth- and BPD-related Obstructive Lung Disease
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Bronchoalveolar lavage (BAL) cells, BAL fluid, bronchial biopsies, airway epithelial brushings, serum, plasma, blood cells, and urine are collected and stored.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Very/extremely prematurely born with BPD: Very/extremely prematurely born (gestational age [GA]< 32 weeks) with bronchopulmonary dysplasia (BPD) as defined by Jobe and Bancalari 2001, age 18-23 years
- Very/extremely prematurely born without BPD: Very/extremely prematurely born (GA< 32 weeks) without BPD in the neonatal period, age 18-23 years
- Asthma full-term control group: Subjects with mild atopic asthma, born at term (GA> 37 weeks), age 18-23 years
- Healthy full-term control group: Healthy participants, born at term (GA>37 weeks), age 18-23 years

SUMMARY:
Obstructive lung disease is an increasing global health problem of pandemic proportions, with COPD alone affecting >10% of the population. Smoking is the main and most well studies risk factor for developing COPD. However, chronic airway obstruction also in never-smoking populations has recently been recognized as an increasing health problem. Prematurely born children, particularly survivors of bronchopulmonary dysplasia (BPD), defined as the need for oxygen therapy up to the 28th day of life for children born prior to gestational week 32, have an increased incidence of both airway obstruction and hyper-reactivity, both representing major risk factors for developing COPD, or asthma, later in life. The purpose of this study is to perform in-depth clinical and molecular characterizations of of the lungs of survivors of BPD as they enter adulthood, and compare these profiles to relevant control groups (individuals with mild asthma, healthy prematurely born, and healthy individuals born at full term). Specifically, alterations at the epigenetic, mRNA, microRNA, protein and metabolite level as well as associated molecular pathways critical in the pathological mechanisms of obstructive lung disease related to premature birth and BPD will be identified.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) is an umbrella diagnosis defined by obstructive lung function impairments, and is likely to be caused by a multitude of etiologies including environmental exposures, genetic predispositions and developmental factors. Due to the heterogeneity of the disease, molecular and mechanistic sub-phenotyping of COPD represents an essential step to facilitate the development of relevant diagnostic and treatment options for this constantly growing patient group. Obstructive lung disease is an increasing global health problem of pandemic proportions, with COPD alone affecting >10% of the population, and predicted by WHO to become the 5th leading cause of morbidity and disability worldwide by year 2020. Smoking is the main and most well studies risk factor for developing COPD. However, chronic airway obstruction also in never-smoking populations has recently been recognized as an increasing health problem: An estimated 10% of patient diagnosed with COPD have never smoked, representing 1% of the general public. Low birth weight and premature birth represent important risk factors for developing pulmonary obstruction in adulthood. Particularly prematurely born children with bronchopulmonary dysplasia (BPD), defined as the need for oxygen therapy up to the 28th day of life for children born prior to gestational week 32, have an increased incidence of both airway obstruction and hyper-reactivity, both representing major risk factors for developing COPD, or asthma, later in life. The purpose of the LUNAPRE study is to perform in-depth clinical and molecular characterizations of of the lungs of survivors of BPD as they enter adulthood, and compare these profiles to relevant control groups. The study encompasses profiling of epigenetic alterations, mRNA, miRNA, proteomes, metabolomes and lipid mediators from multiple lung compartments (airway epithelium, alveolar macrophages, exosomes, and bronchoalveolar exudates) using a range of 'omics platforms, in combination with extensive clinical phenotyping of very prematurely born subjects with- and without BPD in the neonatal period as they enter adulthood, as well as healthy subjects with mild asthma born at term. The primary objective of the study is to identify molecular alterations that persist into adulthood that are related to early onset obstructive lung disease, specifically by correlating clinical phenotypes with multi-molecular 'omics profiling from several lung compartments of the study groups. Secondary goals involve identification of subsets of prognostic/diagnostic biomarkers for classification of the defined subgroups, as well as relevant pharmaceutical targets.

ELIGIBILITY:
Inclusion Criteria:

* Spirometry of postbronchodilator forced expiratory volume in 1 second (FEV1) >50% of predicted level for premature groups

Exclusion Criteria:

* Smoking
* Other lung diseases
* Received antibiotics in the 3 months prior to study entry
* Treatment with oral or inhaled glucocorticoids within past 3 months prior to study entry

Ages: 18 Years to 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants from the two prematurely born groups are recruited from cohort sfollowed since birth at Sach's Children's Hospital, Stockholm. Participants in the full term born groups are recruited from the general population through advertisements.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2013-03-01 (Actual); Primary Completion 2016-09-30 (Actual); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
Forced expiratory volume in 1 second (FEV1) including reversibilityForced expiratory volume in 1 second (FEV1) including reversibilityForced expiratory volume in 1 second (FEV1) including reversibility | Measured at baseline
Forced Vital Capacity (FVC) including reversibility | Measured at baseline
Impulse oscillometry | Measured at baseline
Airway hyper-reactivity (methacholine test) | Measured at baseline
Emphysema and airway wall thickness, as shown on low radiation chest CT scan | Measured at baseline

SECONDARY OUTCOMES:
COPD status (according to GOLD initiative standards as well as LLN) | Determined at baseline
Molecular alterations due to BPD and/or premature birth persisting into adulthood | Determined at baseline
Molecular gender differences | Determined at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Magnus Skold, MD, PhD, Principal Investigator — Karolinska Institute, Karolinska University Hospital; Asa M Wheelock, PhD, Principal Investigator — Karolinska Institutet; Erik Melén, MD, PhD, Principal Investigator — Karolinska Institute, Stockholm Southern General Hospital; Eva Berggren-Brostrom, MD, PhD, Principal Investigator — Stockholm Southern General Hospital; Anders Lindén, MD, PhD, Principal Investigator — Karolinska Institute, Karolinska University Hospital; Sven Nyrén, MD, PhD, Principal Investigator — Karolinska Institute, Karolinska University Hospital; Craig E Wheelock, PhD, Principal Investigator — Karolinska Institutet; Maria J Eriksson, MD, PhD, Principal Investigator — Karolinska Institute, Karolinska University Hospital
Locations (2):
- Sweden (2):
  - Karolinska Institutet/Karolinska University Hospital Solna, Stockholm, Sverige
  - Stockholm Southern General Hospital, Stockholm

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brostrom EB, Thunqvist P, Adenfelt G, Borling E, Katz-Salamon M. Obstructive lung disease in children with mild to severe BPD. Respir Med. 2010 Mar;104(3):362-70. doi: 10.1016/j.rmed.2009.10.008. Epub 2009 Nov 10. PMID 19906521
- [Result] Um-Bergstrom P, Hallberg J, Pourbazargan M, Berggren-Brostrom E, Ferrara G, Eriksson MJ, Nyren S, Gao J, Lilja G, Linden A, Wheelock AM, Melen E, Skold CM. Pulmonary outcomes in adults with a history of Bronchopulmonary Dysplasia differ from patients with asthma. Respir Res. 2019 May 24;20(1):102. doi: 10.1186/s12931-019-1075-1. PMID 31126291
- [Result] Um-Bergstrom P, Pourbazargan M, Brundin B, Strom M, Ezerskyte M, Gao J, Berggren Brostrom E, Melen E, Wheelock AM, Linden A, Skold CM. Increased cytotoxic T-cells in the airways of adults with former bronchopulmonary dysplasia. Eur Respir J. 2022 Sep 29;60(3):2102531. doi: 10.1183/13993003.02531-2021. Print 2022 Sep. PMID 35210327